CLINICAL TRIAL: NCT02362815
Title: Fluid Intake During Labour, Ultrasound Evaluation
Brief Title: Ultrasound Assessment of Clear Liquid Intake During Labour
Acronym: EGTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/27
Record Dates: First submitted 2014-12-26; First posted 2015-02-13 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apple juice (Active Comparator): Patient are allowed to drink up to 400 ml of apple juice
  Interventions: Other: Apple juice
- Control (No Intervention): Patient are not allowed to drink

INTERVENTIONS:
Other: Apple juice — Intervention consists in allowing drinks during labour
  Arms: Apple juice

SUMMARY:
We designed a two arms prospective, randomised, simple blinded trial to compare the impact of clear liquid intake on gastric content before delivery. We hypothesize that there will be no difference between the two groups, leading to safety of clear liquid intake during labour.

DETAILED DESCRIPTION:
Gastric emptying is a major concern for anesthetists in obstetric. In order to prevent the risk of gastric aspiration, we are used to forbid to eat and to drink during labour.

However, this behaviour is controversial and some studies have shown that clear liquid intake can be safe during labour. Informations from a bedside ultrasound examination of the stomach content may be a useful tool to balance benefits and risks of such attitude. This technique has recently been shown very promising in pregnant women for the assessment of the gastric volume.

ELIGIBILITY:
Inclusion Criteria:

* Any pregnant woman at term

Exclusion Criteria:

* Pathologic pregnancy
* Twin pregnancy
* Body mass index above 35 kg/m2 before pregnancy
* Cervix dilation above 8 cm
* Refusal

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Percentage of parturients with a full stomach | average of 6 hours
  A full stomach is defined by an antral area above 300 mm2 evaluated by ultrasound imaging

SECONDARY OUTCOMES:
Parturient comfort | average of 6 hours
  Comfort is evaluated using Labour Agentry Scale
Evolution of the antral area | average of 6 hours
  Antral area are measured by gastric ultrasonography at the beginning and at the end of labour
Anxiety | average of 6 hours
  Anxiety is measured by a Visual Analogic Scale
Pain intensity | average of 6 hours
  Pain is measured by a Visual Analogic Scale

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - CHI Andre Gregoire, Montreuil
  - Tenon, Paris, Île-de-France Region

REFERENCES:
- [Derived] Rousset J, Clariot S, Tounou F, Burey J, Hafiani EM, Feliot E, Quesnel C, Bonnet F, Fischler M. Oral fluid intake during the first stage of labour: A randomised trial. Eur J Anaesthesiol. 2020 Sep;37(9):810-817. doi: 10.1097/EJA.0000000000001278. PMID 32769506